CLINICAL TRIAL: NCT00066339
Title: An IDBBC Single Arm Phase II Trial Evaluating The Activity Of Iressa (ZD1839) In Metastatic Breast Cancer Patients Pretreated With An Antiestrogen And A Non-Steroidal Aromatase Inhibitor (Anastrozole Or Letrozole)
Brief Title: Gefitinib in Treating Patients With Metastatic Breast Cancer That Has Progressed After Antiestrogen and Nonsteroidal Aromatase Inhibitor Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: EORTC-10012; EORTC-10012; IDBBC-10012
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gefitinib

INTERVENTIONS:
Drug: gefitinib

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth.

PURPOSE: Phase II trial to study the effectiveness of gefitinib in treating patients who have metastatic breast cancer that has not responded to antiestrogen and nonsteroidal aromatase inhibitor therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical benefit rate, defined as complete response, partial response, or stable disease after at least 24 weeks, in patients receiving gefitinib for metastatic breast cancer who progressed after prior antiestrogen and nonsteroidal aromatase inhibitor therapy.
* Determine the best overall response rate of patients treated with this drug.
* Determine the progression-free survival of patients treated with this drug.
* Determine the duration of response in patients treated with this drug.
* Determine the safety of this drug in these patients.

OUTLINE: This is a nonrandomized, open-label, multicenter study.

Patients receive oral gefitinib once daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients who go off study in the absence of disease progression are followed every 8 weeks until disease progression.

PROJECTED ACCRUAL: A total of 44 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer
* Radiological and/or clinical evidence of metastatic disease
* Progressive disease after prior therapy with an antiestrogen (e.g., tamoxifen or faslodex) and a nonsteroidal aromatase inhibitor (e.g., anastrozole or letrozole) in the adjuvant and/or metastatic setting* NOTE: *Endocrine therapy must be the last treatment before study entry
* Unidimensionally measurable disease
* No rapidly progressive visceral metastases
* No uncontrolled CNS metastases
* Hormone receptor status:

  * Estrogen receptor and/or progesterone receptor positive

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Not specified

Menopausal status

* Postmenopausal, defined as any of the following:

  * Natural menopause with at least 1 year since last menses
  * Radiation-induced oophorectomy with last menses more than 1 year ago
  * Chemotherapy-induced menopause with 1 year since last menses and serum follicle-stimulating hormone, luteinizing hormone, and plasma estradiol levels in the postmenopausal range
  * Surgical castration

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Transaminases no greater than 2.5 times ULN
* No severe or uncontrolled hepatic disease

Renal

* No severe or uncontrolled renal disease

Cardiovascular

* No severe or uncontrolled cardiac disease

Pulmonary

* No severe or uncontrolled respiratory disease
* No evidence of clinically active interstitial lung disease

  * Asymptomatic chronic stable radiographic changes allowed

Other

* No other malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix, contralateral breast cancer, or nonmelanoma skin cancer
* No psychological, familial, sociological, or geographical condition that would preclude study compliance and follow-up
* No other severe or uncontrolled systemic disease
* No known hypersensitivity to any excipients of gefitinib
* No unresolved chronic toxicity greater than grade 2

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent biologic agents

Chemotherapy

* No more than 1 prior chemotherapy regimen for metastatic breast cancer
* No concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* No concurrent hormonal therapy

Radiotherapy

* Prior radiotherapy allowed
* No concurrent radiotherapy to any metastatic site

Surgery

* No surgery within 4 days after study drug administration

Other

* No prior epidermal growth factor receptor inhibitor therapy
* More than 30 days since prior investigational drugs
* No concurrent use of any of the following:

  * Phenytoin
  * Carbamazepine
  * Rifampin
  * Phenobarbital
  * Hypericum perforatum (St. John's Wort)
* No concurrent systemic retinoids
* No other concurrent investigational drugs or treatments
* No other concurrent anticancer treatments
* Concurrent bisphosphonates for the treatment and prevention of bony metastases are allowed provided therapy was initiated before study enrollment* NOTE: *Bisphosphonates may be initiated during study participation for the treatment of hypercalcemia only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2003-05; Primary Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martine J. Piccart-Gebhart, MD, PhD, Study Chair — Jules Bordet Institute
Locations (1):
- Institut Jules Bordet, Brussels, Belgium